CLINICAL TRIAL: NCT01590251
Title: Yoga for Pain and Opioid Dependence
Acronym: Yoga
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1111009292
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Pain; Opioid Addiction
Keywords: Pain; Addiction; Buprenorphine; Counseling; Methadone; Yoga
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Pain; Behavior, Addictive | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): Gentle yoga for chronic pain and opioid dependence
  Interventions: Other: Yoga
- Educational Counseling (Active Comparator): Educational counseling is a didactic, lecture-discussion format to supplement the information and advice provided in opioid agonist maintenance treatment.
  Interventions: Behavioral: Educational Counseling

INTERVENTIONS:
Other: Yoga — Two yoga sessions per week for 8 weeks (one yoga session is instructional, the other is a practice session.
  Arms: Yoga
Behavioral: Educational Counseling — One didactic session per week of approximately 50 minutes that provides information about chronic pain and substance abuse disorders.
  Arms: Educational Counseling

SUMMARY:
This study is designed to develop an effective adjunctive treatment using yoga for chronic pain and opioid dependence.

DETAILED DESCRIPTION:
This study aims to develop an adjunctive novel treatment intervention using yoga in opioid agonist maintained patients to effectively treat the co-occurring disorders of non-malignant chronic pain and opioid dependence (POD).

Specific Aims:

1) To conduct a pre-pilot phase with 8 patients with POD receiving opioid agonist maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Prescription opioid addiction or heroin addiction
* Moderate to severe chronic pain,
* Understands English

Exclusion Criteria:

* Current suicide or homicide risk
* Life threatening or unstable medical condition
* Medical or psychiatric condition that is judged to be of clinical concern by the PI or admitting clinician
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 8 weeks
  Pain reduction will be measured by patient self-report using standard pain rating scales.
Reduce illicit opioid use | 8 weeks
  Reduced illicit opioid use will be measured by patient self-report and urinalysis testing.

CONTACTS AND LOCATIONS:
Overall Officials: Declan T Barry, Ph.D., Principal Investigator — Yale University
Locations (1):
- MRU, New Haven, Connecticut, United States